CLINICAL TRIAL: NCT06200064
Title: Comparative Effect of Post Isometric Relaxation and Self-stretching on Non-specific Neck Pain in Working Age Persons
Brief Title: Physiotherapy for Non-specific Neck Pain in Working Age Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Principal Investigator, Vilma Dudoniene, Lithuanian Sports University, Lithuanian Sports University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LithuanianSportsU-19
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain; Non-specific Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This study is a four week, single blinded randomized controlled trial with pre-post design comparing self-stretching exercise group with post-isometric relaxation exercise group.
Who Masked: Outcomes Assessor
Masking Description: outcomes were measured by separate physiotherapist, who did not provide prescribed intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-stretching exercise group (Experimental): Static neck muscle self-stretching exercises were performed for 30 min. after the TENS procedure. Every muscle in the neck region (head rotator cuff, neck stair muscles, upper part of the trapezius muscle, scapula levator muscle, semiscapular neck muscle, upper oblique head muscle, girdle head and neck muscles, and deep anterior neck flexor muscles) were stretched 3 times for 30 seconds per muscle group. While performing exercises, the subjects applied resistance with their hands. All exercises were performed without causing pain.
  Interventions: Other: Self-stretching exercise group
- Post-isometric relaxation exercise group (Experimental): The investigators used one of the autogenic inhibition techniques - post-isometric relaxation (PIR), known as the muscle "contraction-relaxation" technique, during which, the subject is lying on his back, he is asked to press his head in the specified direction (50% of the subject's maximum pressure force). to the resistance provided by the therapist. During the press, resistance was provided for 10 seconds and followed by a passive stretch of the muscle in the opposite direction of movement. A total of 5 repetitions are performed for each muscle with a 5-second break. All movements are performed without causing pain of more than moderate intensity.
  Interventions: Other: Post-isometric relaxation exercise group

INTERVENTIONS:
Other: Self-stretching exercise group — Static neck muscle self-stretching exercises were performed for 30 min. after the TENS procedure. Every muscle in the neck region (head rotator cuff, neck stair muscles, upper part of the trapezius muscle, scapula levator muscle, semiscapular neck muscle, upper oblique head muscle, girdle head and neck muscles, and deep anterior neck flexor muscles) were stretched 3 times for 30 seconds per muscle group. While performing exercises, the subjects applied resistance with their hands. All exercises were performed without causing pain.
  Arms: Self-stretching exercise group
Other: Post-isometric relaxation exercise group — The investigators used one of the autogenic inhibition techniques - post-isometric relaxation (PIR), known as the muscle "contraction-relaxation" technique, during which, the subject is lying on his back, he is asked to press his head in the specified direction (50% of the subject's maximum pressure force). to the resistance provided by the therapist. During the press, resistance was provided for 10 seconds and followed by a passive stretch of the muscle in the opposite direction of movement. A total of 5 repetitions are performed for each muscle with a 5-second break. All movements are performed without causing pain of more than moderate intensity.
  Arms: Post-isometric relaxation exercise group

SUMMARY:
The goal of this clinical trial is to learn about the effects of two different physiotherapy methods on non-specific neck pain in working age individuals. The main questions it aims to answer are:

* What is the effect of self stretching exercise on non-specific neck pain, functional disability, range of motion of the cervical spine and hand muscle strength in working age individuals?
* What is the effect of post-isometric relaxation exercise on non-specific neck pain, functional disability, range of motion of the cervical spine and hand muscle strength in working age individuals?
* Is any of the applied interventions (self-stretching or post-isometric relaxation exercise) superior to each other?

Participants will:

* be evaluated by an experienced physiotherapist who will perform the interview and physical examination. Interview includes questions about the age, sex, work profile, pain intensity and duration, and other complaints. Physiotherapy examination includes a range of motion measurement, hand grip muscle strength and functional disability index evaluation.
* Two different interventions will be prescribed to the randomly assigned study participants: post-isometric relaxation and self-stretching. Duration of interventions for both groups is 4 weeks (3 times per week, 12 sessions). Duration of one session - 45 min.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the effects of two different physiotherapy methods on non-specific neck pain in working age individuals. The main questions it aims to answer are:

What is the effect of self stretching exercise on non-specific neck pain, functional disability, range of motion of the cervical spine and hand muscle strength in working age individuals? What is the effect of post-isometric relaxation exercise on non-specific neck pain, functional disability, range of motion of the cervical spine and hand muscle strength in working age individuals? Is any of the applied interventions (self-stretching or post-isometric relaxation exercise) superior to each other?

Participants will:

be evaluated by an experienced physiotherapist who will perform the interview and physical examination. Interview includes questions about the age, sex, work profile, pain intensity and duration, and other complaints. Physiotherapy examination includes a range of motion measurement, hand grip muscle strength and functional disability index evaluation.

Two different interventions will be prescribed to the randomly assigned study participants: post-isometric relaxation and self-stretching. Duration of interventions for both groups is 4 weeks (3 times per week, 12 sessions). Duration of one session - 45 min.

ELIGIBILITY:
Inclusion Criteria:

* current neck pain,
* neck pain duration for at least 12 weeks,
* admission through outpatient clinic in Lithuania.

Exclusion Criteria:

* neurological disorders related to neck pain,
* red flags (night pain, severe muscle spasm, loss of involuntary weight, symptom mismatch),
* previous neck surgery,
* low back pain,
* medications used for pain.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from Baseline Quality of Life at 4 weeks
  Neck pain intensity was assessed using a visual analogue scale (VAS) on a 10-cm line with end-point descriptors such as 'no pain' marked at the left end and 'worst pain imaginable' marked at the right end. Patients were asked to mark a point on the line that best represented their pain at the time of the evaluation. The distance from 'no pain' to the patient's mark was then measured and recorded as the VAS score: 0 cm was defined as no pain, 1-3 cm as mild pain, 4 or 5 cm as moderate pain, 6-8 cm as severe pain and 9 or 10 cm as the worst pain imaginable.

SECONDARY OUTCOMES:
Cervical spine range of motion | Change from Baseline Quality of Life at 4 weeks
  ROM was measured using bubble inclinometer, which was placed on the top of the patient's head, along the sagittal plane to measure neck flexion and extension, when the patient was in sitting position. Side bending was measured from the same starting position just as the inclinometer was placed in the frontal plane on the top of the patient's head. Rotations to the left and right were taken from the supine position with an inclinometer placed on the forehead. The inclinometer's reading at the starting position was 0. The readings of ROM were taken when the end point of movement was reached. In our study, three repetitions were performed in each direction, and the average value was taken for analysis.
Hand grip strength | Change from Baseline Quality of Life at 4 weeks
  Hand grip strength was measured using a hand dynamometer (Saehan SH5001, Germany). Grip strength of the dominant and non-dominant hand was measured when seated with the shoulder neutrally rotated and adducted, the elbow flexed at 90°, and the wrist and forearm in a neutral position. The maximum grip strength was measured in kilograms (kg). Three measurements were taken with 60 s rest between each trial and the average result was recorded.
The Neck Disability Index | Change from Baseline Quality of Life at 4 weeks
  The Neck Disability Index (NDI) questionnaire consists of 10 items. Each item on the scale is scored from 0 to 5, where all the scores are added to total points and interpreted as percentages i.e., 0 point or 0% means no activity limitation, and 50 points or 100% means complete activity limitation. The NDI is a reliable and valid questionnaire in neck pain patients with intraclass correlation ranges between 0.50-0.98. Patients scored between 0-4 points (0-8%) are considered with no disability, between 5-14 points (10-28%) with mild disability, 15-24 points (30-48%) - moderate disability, 25-34 points (50- 64%) - severe disability, and 35-50 points (70-100%) - complete disability

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Dudoniene, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No